CLINICAL TRIAL: NCT01289886
Title: BR-A-657, A Phase 1, Double-blind, Placebo-controlled, Ascending Single Oral Dose Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Male Subjects Incorporating a Comparison of Fed/Fasted Pharmacokinetics
Brief Title: Fimasartan (BR-A-657) Single Oral Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Covance (Industry)
Responsible Party: Paik, Assistant manager, Boryung Pharm. Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2290/2
Record Dates: First submitted 2010-12-13; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-01

CONDITIONS: Essential Hypertension
Keywords: single-dose; pharmacokinetic; pharmacodynamic; safety
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A (Other): BR-A-657 20mg or placebo
  Interventions: Drug: BR-A-657
- Arm B (Other): BR-A-657 60mg or placebo
  Interventions: Drug: BR-A-657
- Arm C (Other): BR-A-657 120mg or placebo
  Interventions: Drug: BR-A-657
- Arm D (Other): BR-A-657 240mg or placebo
  Interventions: Drug: BR-A-657
- Arm E (Other): BR-A-657 480mg or placebo
  Interventions: Drug: BR-A-657

INTERVENTIONS:
Drug: BR-A-657 — 20, 60, 120, 240, 360, 480mg or placebo tablet
  Other Names: Fimasartan; 20, 60, 120, 240, 360, 480mg

SUMMARY:
The objective of this study is to determine the safety and tolerability and to determine the Pharmacokinetic and Pharmacodynamic (PK/PD) of ascending single oral dose of BR-A-657 in healthy male subjects.

DETAILED DESCRIPTION:
BR-A-657 20, 50, 120, 240, 360, 480mg or placebo were administered once to healthy male subjects.

Pharmacokinetic and Pharmacodynamic(PK/PD) parameters were monitored at pre-specified times from each subjects.

PK parameters: Area Under the Curve(AUC), Cmax, half-life, etc. PD parameters: Aldosterone, Plasma renin activity, Angiotensin I, Angiotensin II Adverse events are reported.

ELIGIBILITY:
Inclusion Criteria:

* male of 18-55 years old
* Body Mass Index(BMI) 19-29kg/m2
* subjects in good health
* subjects with written informed consent

Exclusion Criteria:

* subjects with multiple drug allergy or allergy to Angiotensin Receptor Blocker(ARB)
* subjects with medication that affect drug absorption or elimination within 30days.
* subjects with orthostatic hypotension of >20mmHg decrease of Systolic Blood Pressure(SBP)
* subjects with history of neurologic, liver, renal, gastrointestinal, cardiovascular, psychological or other major disorder

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2003-11 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
No of subjects with Adverse events(AE) from each observations | up to 5~7days post-dose
  1. AE reporting: Pre dose, 3, 12, 24h, (48 h: Groups C, D, E) post dose
  2. Vital signs: Pre dose*, 0.5, 1*, 2, 4*, 6, 8*, 12 and 24* h post dose (*:both supine and standing)
  3. ECG: Pre dose, 2, 4, 8 and 24 h post dose
  4. Clinical laboratory examination: Pre dose and 24 h post dose
  5. Physical examination: predose, 5~7days post dose
  6. Body weight: predose, 5~7days post dose

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUC) | 0.5,1,1.5,2,3,4,6,8,12,16,24,(48: Groups C, D, E)h
Maximum observed plasma concentration (Cmax) | 0.5,1,1.5,2,3,4,6,8,12,16,24,(48: Groups C, D, E)h
Time of the maximum observed plasma concentration (Tmax) | 0.5,1,1.5,2,3,4,6,8,12,16,24,(48: Groups C, D, E)h
Apparent total plasma clearance (CL/F) | 0.5,1,1.5,2,3,4,6,8,12,16,24,(48: Groups C, D, E)h
Apparent plasma terminal elimination half life (t½) | 0.5,1,1.5,2,3,4,6,8,12,16,24,(48: Groups C, D, E)h

CONTACTS AND LOCATIONS:
Overall Officials: E Engmann, MB ChB, Principal Investigator — Covance Clinical Research Unit